CLINICAL TRIAL: NCT03911947
Title: Assessing the Ventilatory Parameters in Patients With Acute Respiratory Failure After Vibroacoustic Pulmonary Therapy.
Brief Title: Evaluation of the Effectiveness of Vibroacoustic Therapy in the Complex Treatment of Acute Respiratory Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Astana Medical University (Other)
Responsible Party: Principal Investigator, Aidos Konkayev, Chair of department, Astana Medical University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1972
Record Dates: First submitted 2019-04-08; First posted 2019-04-11 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Respiratory Failure
Keywords: Vibroacoustic therapy, acute respiratory failure, pneumonia
MeSH Terms: conditions — Respiratory Insufficiency; Pneumonia

STUDY DESIGN:
Intervention Model Description: monitoring of treatment of patients with respiratory failure, the list of therapeutic measures which includes vibroacoustic therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SaO2 (oxygen status) (Active Comparator): Measurment 4 times per day, ABA (acid-bases analyses)
  Interventions: Device: Vibrolung
- PaO2/FiO2 (respiratory index) (Active Comparator): Measurment 4 times per day, ABA (acid-bases analyses)
  Interventions: Device: Vibrolung
- AB (actual bicarbonat level) (Active Comparator): Measurment 4 times per day, ABA (acid-bases analyses)
  Interventions: Device: Vibrolung

INTERVENTIONS:
Device: Vibrolung — Device for vibroacoustic respiratory therapy

SUMMARY:
Evaluation of the effectiveness of vibroacoustic therapy in the complex treatment of acute respiratory failure

DETAILED DESCRIPTION:
Assessing the dynamics of changes in physical, instrumental and laboratory parameters in patients with acute respiratory failure taken in the study according to the inclusion criteria and comparing the results with the control group, studying the effectiveness of vibroacoustic lung therapy.

ELIGIBILITY:
Inclusion Criteria:

* adults
* P/F less 300 torr
* ARDS by Berlin convention

Exclusion Criteria:

* children
* acute stroke
* acute coronary syndrome
* DVT
* implanted pacemaker
* rib fracture
* infection on chest

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Change of time spent on ventilation | 1-2 days
  Changing of the time spent by patients on mechanical ventilation

CONTACTS AND LOCATIONS:
Locations (5):
- Kazakhstan (5):
  - City clinical hospital №7, Almaty
  - City clinical hospital №1, Astana
  - National Cardiac Surgery Center, Astana
  - Scientific Research Institute of Traumatology and Orthopedics, Astana
  - Regional cardiology center, Shymkent

IPD SHARING:
Plan to Share IPD: No